CLINICAL TRIAL: NCT02378948
Title: Nutritional Route in Esophageal Resection Trial II (NUTRIENT II): a Randomized Controlled Trial
Brief Title: Nutritional Route In Esophageal Resection Trial II
Acronym: NUTRIENTII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Misha D.P. Luyer, MD, PhD, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL52591.060.15
Record Dates: First submitted 2015-02-23; First posted 2015-03-04 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Neoplasms
Keywords: Esophagectomy; Nutrition; Oral feeding; Enteral feeding; Pulmonary complications; Anastomotic leakage; Quality of life
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early oral feeding (Experimental): Liquid oral feeding directly after esophagectomy.
  Interventions: Dietary Supplement: Liquid oral feeding
- Delayed oral feeding (No Intervention): Liquid oral feeding 5 days after esophagectomy

INTERVENTIONS:
Dietary Supplement: Liquid oral feeding — Liquid oral feeding (water, soup, porridge, nutritional supplements etc.)
  Arms: Early oral feeding

SUMMARY:
The aim of this study is to investigate the effects of early start versus delayed start of oral intake on postoperative functional recovery after an esophagectomy.

DETAILED DESCRIPTION:
Early oral feeding is safe and beneficial in most types of gastro-intestinal surgery and is a crucial part of fast track or enhanced recovery protocols. Following esophagectomy, fast track programs are increasingly being applied, resulting in a reduced length of stay, perioperative morbidity and hospital charges. In a previous feasibility study (Nutrient I trial) has been shown that direct oral intake following esophagectomy was feasible and did not result in an increase of major complications. It remains unclear what the best strategy is for nutrition in the early postoperative phase following esophagectomy. The aim of this study is to investigate the effects of early start versus delayed start of oral intake on postoperative recovery and pulmonary complications following esophagectomy.

Patients will be recruited at the outpatient clinic of the Catharina Hospital Eindhoven and the Hospital Group Twente.Patients will enroll in the early oral feeding group or the delayed oral feeding group. The early oral feeding group will receive liquid oral nutrition directly after surgery. Patients in the delayed oral feeding group will receive enteral tube feeding (via a jejunostomy) for 5-7 days (standard protocol in The Netherlands). After these 5-7 days a liquid oral diet is initiated.

Patient characteristics and clinical parameters are registered in an electronic database. All surgical complications are classified using the Clavien-Dindo classification15 (Appendix II). An independent investigator will check functional recovery daily. Data is provided by local investigator via an online checklist (electronic case report form / website). Quality of life and Symptoms are scored using the European organization for research and treatment of cancer questionnaire (QLQ-C30/EORTC-OG25)16 at baseline (5 weeks after neoadjuvant treatment), 6 weeks, 3 months and 6 months postoperatively. Cost-effectiveness is scored via EQ-5D-5L, iMTA Medical Consumption Questionnaire (iMCQ) and Productivity Cost Questionnaire (iPCQ). Nutritional status will be measured using the actual caloric and protein intake versus the needed caloric and protein intake. Long-term outcome parameters such as local recurrence, overall and cancer-specific survival will be registered in a database until the end of the study.

The sample size calculation is based on functional recovery as primary outcome. Functional recovery is the time to surgical recovery according to the definition described previously. Patients in our historic cohort (1 week artificial nutrition) were at least considered functional recovered by a mean of 12 days post-surgery. Patients in the NUTRIENT I were at least functional recovered at day 10 postoperative (mean) following an esophagectomy. In this trial we consider a reduction of 2 days in functional recovery as clinically significant. Using a Power of 80%, an alpha of 5% and a standard deviation of 4 days, a total of 128 patients (64 patients in each group) is needed to show this difference. It is expected that the primary outcome will not be normally divided and therefore an extra 15% inclusion is necessary, requiring a total of 148 patients (74 patients in each group). Interim-analyses will be performed following 50 and 100 patients and will be checked by an independent physician.

All analyses will be done according to the intention-to-treat approach in which all randomized patients are included, regardless of adherence to study protocol. Occurrences of the primary and secondary endpoints are compared between the treatment groups. Results are presented as risk ratios with corresponding 95% confidence intervals. A two-tailed P < 0.05 is considered statistically significant. To compare the groups the data will be tested for normal distribution and an unpaired T-test will be performed when appropriate, otherwise the Mann-Whitney U or Chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients that undergo a (minimally invasive) esophagectomy with intrathoracic anastomosis.
* written informed consent
* age >18 years

Exclusion Criteria:

* Inability for oral intake
* Inability to place a surgical feeding jejunostomy
* Mental retardation
* Swallowing disorder
* Achalasia
* Malnutrition (defined as >15% weight loss just before start of the surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Functional recovery | up to 4 weeks after surgery
  The primary outcome parameter is the day of functional recovery. Functional recovery is defined as postoperative patients who are free of IV fluid, have adequate pain control, restoration of mobility to an independent level, have sufficient caloric intake and no signs of active infection.

SECONDARY OUTCOMES:
Pulmonary complications | up to 4 weeks after surgery
  (Pneumonia, Acute respiratory distress syndrome, respiratory insufficiency requiring treatment)
Anastomotic leakage | up to 4 weeks after surgery
Nutritional status (weight loss, intake) | postoperative day 2, 5 and 14
Need for parenteral feeding/ placement of a nasojejunal feeding tube | up to 2 weeks after surgery
Need for additional surgical, radiological or endoscopic interventions | up to 4 weeks after surgery
30-day surgical complications (classified according to Clavien-Dindo) | up to 4 weeks after surgery
  classified according to Clavien-Dindo
Other complications requiring treatment | up to 4 weeks after surgery
  i.e. urinary tract infection
Need for ICU admission and total length of ICU stay | up to 4 weeks after surgery
Quality of life | 6 weeks after neoadjuvant treatment, 6 weeks, 3 months en 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Misha DP Luyer, MD, PhD, Study Chair — Catharina Ziekenhuis Eindhoven
Locations (2):
- Netherlands (2):
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant
  - Ziekenhuisgroep Twente, Almelo, Overijssel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berkelmans GH, Wilts BJ, Kouwenhoven EA, Kumagai K, Nilsson M, Weijs TJ, Nieuwenhuijzen GA, van Det MJ, Luyer MD. Nutritional route in oesophageal resection trial II (NUTRIENT II): study protocol for a multicentre open-label randomised controlled trial. BMJ Open. 2016 Aug 5;6(8):e011979. doi: 10.1136/bmjopen-2016-011979. PMID 27496239